CLINICAL TRIAL: NCT03720613
Title: Risk of Major Adverse Cardiovascular Events Among Users of Naldemedine Compared With Other Medications Used for Opioid Induced Constipation in Adult Patients With Chronic Non-Cancer Pain in a Healthcare Claims Database
Brief Title: Risk of Major Adverse Cardiovascular Events for Naldemedine & Other Medications for Opioid Induced Constipation
Status: Recruiting | Type: Observational
Sponsor: BioDelivery Sciences International (Industry)
Collaborators: HealthCore, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1711V9241
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Opioid-induced Constipation
Keywords: naloxegol; major adverse cardiovascular event (MACE); opioid induced constipation (OIC); lubiprostone; naldemedine
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naldemedine; Lubiprostone; naloxegol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Naldemedine: Patients with chronic non-cancer pain who initiated naldemedine treatment for opioid-induced constipation.
  Interventions: Drug: Naldemedine
- Lubiprostone: Patients with chronic non-cancer pain who initiated lubiprostone treatment for opioid-induced constipation.
  Interventions: Drug: Lubiprostone
- Naloxegol: Patients with chronic non-cancer pain who initiated naloxegol treatment for opioid-induced constipation.
  Interventions: Drug: Naloxegol

INTERVENTIONS:
Drug: Naldemedine — 0.2 mg tablet once a day at any time with or without food
  Other Names: Symproic®
  Groups: Naldemedine
Drug: Lubiprostone — 0.024 mg twice a day [adjust dose based on liver function]
  Other Names: Amitiza®
  Groups: Lubiprostone
Drug: Naloxegol — 25 mg tablet once a day in morning, 1 hour before or 2 hours after food
  Other Names: Movantik®
  Groups: Naloxegol

SUMMARY:
The research objective is to characterize the risk of a major adverse cardiovascular event (MACE) among new users of naldemedine versus new users of lubiprostone and new users of naloxegol as comparator opioid induced constipation (OIC) medications.

DETAILED DESCRIPTION:
This is a prevalent new user cohort study conducted using multiple databases linkable to medical records and the National Death Index (NDI) to assess MACE risk among adult patients with chronic non-cancer pain receiving naldemedine or a comparator OIC medication. The uptake of naldemedine and comparator OIC medications will be monitored for each database annually until a sufficient number of patients to support the comparative analyses in the safety assessment phase is accrued. The safety assessment phase will commence at the conclusion of the monitoring phase.

ELIGIBILITY:
Inclusion Criteria:

* At least one dispensing of naldemedine or lubiprostone or naloxegol without prior use in the database of either medication (index date)
* At least two dispensings of opioids within six months prior to and including the index date, with at least a combined 31 cumulative days supply
* At least 18 years of age or older on the index date
* At least six months of continuous health plan coverage that includes medical and pharmacy benefits prior to and including the index date

Exclusion Criteria:

* Any acute MACE (non-fatal MI or non-fatal stroke) within six months before or on the index date
* Any cancer treatment or cancer pain diagnosis within six months before or on the index date
* Prior use of methylnaltrexone, alvimopan or naloxegol within six months before or on the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include new users of naldemedine or one of the comparator OIC medications (lubiprostone or naloxegol) who satisfy all of the inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 34532 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2030-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Major Adverse Cardiovascular Event | 5 years
  A composite of major adverse cardiovascular events, cardiovascular (CV) death, nonfatal myocardial infarction (MI), and non-fatal stroke; participants with major adverse cardiovascular events will be identified using claims data and the national death index.

SECONDARY OUTCOMES:
Number of Participants with Cardiovascular Death | 5 years
  Cardiovascular death is defined by the underlying cause of death and will include death from acute MI, sudden cardiac death, heart failure, stroke, cardiovascular procedure, cardiovascular hemorrhage, and other cardiovascular causes. Cardiovascular death will be identified using claims data and the national death index.
Number of Participants with Nonfatal Myocardial Infarction | 5 years
  Participants with nonfatal myocardial infarction will be identified using claims data.
Number of Participants with Nonfatal Stroke | 5 years
  Participants with nonfatal stroke will be identified using claims data.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lanes, Principal Investigator — HealthCore, Inc.
Locations (1):
- Research Site, Wilmington, Delaware, United States